CLINICAL TRIAL: NCT00433706
Title: Economic Evaluation of Image Guided Radiation Therapy For Prostate Cancer
Brief Title: Image Guided Radiation Therapy For Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CSET 1248; IGRT-P
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Prostate Cancer
Keywords: Prostate adenocarcinoma treated by radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (2):
- Control position by 3DOBI daily (Experimental)
  Interventions: Procedure: Control position by 3DOBI before the fraction
- Standard imaging (Active Comparator)
  Interventions: Procedure: Standard imaging

INTERVENTIONS:
Procedure: Control position by 3DOBI before the fraction
  Arms: Control position by 3DOBI daily
Procedure: Standard imaging
  Arms: Standard imaging

SUMMARY:
During the 7 to 8 weeks of conformal radiotherapy for prostate carcinoma, the prostate has an intra-pelvic motion which is not detectable by the conventional portal imaging. This prostate motion may lead to a mistargeting, which possibly decreases the local control. On the other hand, the new 3D on board imaging (3D OBI) allows to localize the target but is expensive. The cost/effectiveness ratio is not well established, as well as the frequency of using such imaging during the course of radiation.

ELIGIBILITY:
Inclusion Criteria:

* prostate adenocarcinoma
* intermediate / high risk group
* N0 or N -
* treatment by conformal radiotherapy (including or not IMRT), with or without androgen deprivation

Exclusion Criteria:

* pelvic irradiation
* metal objects in the pelvis

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2007-06; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Prostate position under the LINAC is checked by 3D OBI (mainly cone-beam imaging, CBI) performed before the fraction.
To validate the optimal strategy of IGRT for prostate adenocarcinoma based on 2 and 5 year-disease free survival rates (events= biochemical failure or death).

SECONDARY OUTCOMES:
Rectal and bladder, acute and late toxicities (CTCAE, SOMA-LENT)
Cost comparison and cost/effectiveness analysis
2 and 5 years clinical relapse free survival rates
Lack of dose in the prostate in case of decreasing the CBI frequency (using the 1rst arm for testing)

CONTACTS AND LOCATIONS:
Overall Officials: Renaud DE CREVOISIER, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France